CLINICAL TRIAL: NCT02780453
Title: Prophylactic Negative Pressure Dressings for Closed Laparotomy Wounds - A Randomised, Controlled, Open Label Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of Limerick (Other)
Responsible Party: Principal Investigator, Peter O'Leary, Surgery SPR, University Hospital of Limerick
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PICO Trial
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Negative pressure dressing (Experimental): Negative pressure dressing
  Interventions: Device: Negative pressure dressing
- Standard dressing (Active Comparator): Standard wound dressing
  Interventions: Device: Standard wound dressing

INTERVENTIONS:
Device: Negative pressure dressing
  Arms: Negative pressure dressing
Device: Standard wound dressing
  Arms: Standard dressing

SUMMARY:
Laparotomy wounds are associated with high rates of surgical site infections (SSI). The effect of prophylactic negative pressure dressing of closed incisional wounds on SSI rates is inconclusive.

ELIGIBILITY:
Inclusion Criteria:

* Elective and emergency abdominal surgery

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Surgical site infection rate | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Limerick, Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] O'Leary DP, Peirce C, Anglim B, Burton M, Concannon E, Carter M, Hickey K, Coffey JC. Prophylactic Negative Pressure Dressing Use in Closed Laparotomy Wounds Following Abdominal Operations: A Randomized, Controlled, Open-label Trial: The P.I.C.O. Trial. Ann Surg. 2017 Jun;265(6):1082-1086. doi: 10.1097/SLA.0000000000002098. PMID 27926575